CLINICAL TRIAL: NCT07332702
Title: Detection of Cis Duplications of the SMN1 Gene Using Long-read Analysis to Address a Major Issue in Genetic Counseling for Spinal Muscular Atrophy
Brief Title: Long Read Analysis in Spinal Muscular Atrophy - LOREASI
Acronym: LOREASI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/0154/HP
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy (SMA)
Keywords: SMA, SMN1, long read, cis duplication, genetic counselling
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophy, Type IV | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): subjects carrying 1 or 3 copies of the SMN1 gene and a variable number of copies of the SMN2 gene
  Interventions: Genetic: blood sample
- Test group (Experimental): subjects carrying a 2+0 genotype (two copies of the SMN1 gene in cis on one allele and a deletion on the other allele)
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — For subjects who agree to participate in the study, a blood sample will be taken (2x5 mL on EDTA) and sent the same day at 4°C to the genetics laboratory at Rouen University Hospital using a carrier that guarantees delivery on D+1

SUMMARY:
Spinal Muscular Atrophy (SMA) is a severe neuromuscular disease caused by deletion of the SMN1 gene, with the most severe form leading to death in children without treatment. Genetic counselling to detect couples where both partners are carriers is particularly important. In some countries, preconception screening is offered. However, some carriers escape detection due to the existence of two copies of the SMN1 gene side-by-side (2+0 genotype). Currently, no molecular genetic methods used for diagnostic purposes can detect these 2+0 genotypes, which pose a significant challenge in genetic counselling.

This study aims to use new technologies based on the analysis of ultra-long molecules to detect side-by-side duplications of the SMN1 gene to detect heterozygous subjects not identified by current techniques and improve genetic counselling.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is a severe autosomal recessive neuromuscular disease, with the most severe form leading to death in children without treatment. Genetic counseling to detect couples where both partners are heterozygous is particularly important. In some countries, preconception screening is offered. However, some individuals' heterozygous status escape detection due to the existence of a cis duplication of the SMN1 gene on the second allele ([2+0] genotype). Currently, no molecular genetic methods used for diagnostic purposes can detect these [2+0] genotypes, which poses a significant challenge in genetic counseling.

The SMN1 gene, responsible for SMA, is located in the 5q11q13 region, which remains poorly understood in the human reference genome ("dark region"). The architecture of this inverted duplicated region favors recombination events that lead to deletions, duplications, and gene conversions. The SMN1 gene, located in the telomeric region, has a very homologous copy, the SMN2 gene, located in the centromeric region. The lack of detailed knowledge about duplication events hinders the development of molecular tools aimed at improving genetic counseling.

This study aims to use new technologies based on the analysis of ultra-long molecules to detect cis duplication of the SMN1 gene. We will assess the usefulness of optical mapping (Bionano) to analyze this complex region.

ELIGIBILITY:
Inclusion Criteria

• Adult Subject:

* Subject with either:

  * 1 or 3 copies of the SMN1 gene (control group) and a variable number of copies of the SMN2 gene
  * 2 copies of the SMN1 gene in cis (2+0 genotype) (test group)
* Affiliation to French health insurance
* Signed consent form

Exclusion Criteria

* Pregnant or breastfeeding women
* Individuals deprived of liberty by an administrative or judicial decision, or those under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Ability to identify a [2+0] SMN1 genotype | From enrollment until the end of the analyses (36 months)

SECONDARY OUTCOMES:
Ability to perform assembly of ultra-long molecules of DNA | From enrollment until the end of the analyses (36 months)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rouen, Rouen, France